CLINICAL TRIAL: NCT07126808
Title: Effectiveness of a Simulation-Based Cardiopulmonary Resuscitation Workshop Among University Students at Eastern International University: A Randomized Waitlist-Controlled Trial
Brief Title: Simulation-Based CPR Workshop for University Students at Eastern International University
Acronym: EIU-CPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Hong Liem (Other)
Responsible Party: Sponsor-Investigator, Le Hong Liem, Lecturer, School of Nursing, Eastern International University, Eastern International University
Organization: Eastern International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EasternIU
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Primary Condition/Focus: Cardiopulmonary Resuscitation Training
Keywords: Basic Life Support Training; CPR; BLS training; Cardiopulmonary Resuscitation Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. The intervention group will receive the simulation-based CPR workshop immediately after baseline assessment. The waitlist control group will receive no intervention until after the follow-up assessment, at which point they will receive the same workshop to ensure equitable training for all participants.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group assignments during data collection and scoring to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Simulation-Based CPR Workshop (Experimental): Participants receive a 4-hour simulation-based CPR workshop immediately after baseline. Training follows AHA guidelines and the NLN Jeffries Simulation Framework and includes: pre-briefing; instructor-led demonstration; hands-on practice on manikins (rate, depth, recoil, ventilation, AED use); scenario simulation with team roles; and structured debriefing. Trainer: BLS-certified faculty. Group size ~12-20; trainer:student ≈1:6. Outcomes (skills, knowledge, attitude, self-efficacy) assessed at baseline (T1), immediate post-test (T2), and 3-month follow-up (T3).
  Interventions: Behavioral: Simulation-Based CPR Workshop
- Waitlist Control - Delayed Workshop (No Intervention): Participants follow usual activities during the study period and do not receive the CPR workshop until after the follow-up assessment to ensure equity. They complete the same assessments as the intervention arm at baseline (T1), immediate post-test timing (T2, without training), and 3-month follow-up (T3). After T3 data collection, they receive the identical 4-hour simulation-based CPR workshop (same content, trainers, and format) as the intervention group.

INTERVENTIONS:
Behavioral: Simulation-Based CPR Workshop — A 4-hour, in-person simulation-based cardiopulmonary resuscitation (CPR) workshop designed for non-healthcare university students, following American Heart Association 2020 guidelines and the NLN Jeffries Simulation Framework. The training includes: (1) pre-briefing on OHCA and CPR importance; (2) instructor-led demonstration using manikins; (3) guided hands-on practice with real-time feedback; (4) scenario-based simulation with assigned team roles; and (5) structured debriefing for reflection and feedback. Skills practiced include scene safety, assessing responsiveness, high-quality chest compressions, rescue breathing, AED use, and team communication. Trainer-to-student ratio is approximately 1:6.
  Arms: Intervention - Simulation-Based CPR Workshop

SUMMARY:
This study aims to evaluate the effectiveness of a simulation-based cardiopulmonary resuscitation (CPR) workshop in improving knowledge, practical skills, attitudes, and self-efficacy among university students at Eastern International University, Vietnam. Out-of-hospital cardiac arrest (OHCA) survival rates in Vietnam remain low, partly due to limited bystander CPR and lack of AED use. University students, especially those outside healthcare fields, represent a large and accessible population who could serve as first responders in emergencies.

The workshop is designed according to the NLN Jeffries Simulation Framework and current American Heart Association guidelines. It includes instructor-led demonstrations, hands-on practice using manikins, scenario-based simulations, and structured debriefing. The training focuses on essential CPR steps, AED operation, and teamwork in emergency situations.

This randomized waitlist-controlled trial will assign participants to either an immediate training group or a waitlist control group who will receive the same training after the follow-up phase. Primary outcomes include improvements in CPR skills, measured through a standardized performance checklist. Secondary outcomes include knowledge, self-efficacy, and attitudes toward performing CPR. Assessments will be conducted before, immediately after, and three months after the intervention.

Findings from this study will provide empirical evidence on the impact of simulation-based CPR education for non-healthcare university students in Vietnam. The results could support integrating CPR workshops into university curricula and scaling up community-based emergency response training programs to increase bystander CPR rates and improve OHCA survival.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a serious public health challenge, with low survival rates in many countries, including Vietnam, where bystander CPR is rarely performed, and AEDs are seldom used in public. Previous studies in Vietnam show limited CPR knowledge, skills, and willingness to act among non-healthcare university students. Despite evidence supporting simulation-based CPR education in other countries, no randomized controlled trial has evaluated such an intervention for this population in Vietnam.

This study is a randomized waitlist-controlled trial designed to evaluate a simulation-based CPR workshop for university students at Eastern International University. Participants will be randomly assigned to an intervention group or a waitlist control group. The intervention group will receive the workshop immediately, while the waitlist control group will receive it after the follow-up assessment, ensuring equitable training for all participants.

The workshop, based on the NLN Jeffries Simulation Framework and aligned with American Heart Association guidelines, includes pre-briefing, instructor-led demonstrations, hands-on skill practice with manikins, realistic scenario simulations, and structured debriefing. Training emphasizes high-quality chest compressions, effective ventilations, AED use, scene safety, and teamwork.

Primary outcomes will focus on improvements in CPR skills, assessed using a standardized performance checklist. Secondary outcomes will measure CPR knowledge, attitudes, and self-efficacy using validated instruments. Data will be collected at baseline, immediately post-training, and at three months follow-up. Statistical analyses will include repeated measures ANOVA to assess changes over time and between groups.

By addressing a critical gap in Vietnam's CPR education, this study aims to provide empirical evidence supporting the integration of simulation-based CPR training into non-medical university curricula. If proven effective, the model could be scaled to other educational and community settings, contributing to improved bystander CPR rates and better OHCA survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a student at Eastern International University (EIU).
* Aged 18 years or older.
* Willing to participate in the study and sign the informed consent form.
* Able to communicate and understand Vietnamese.
* Have not participated in a simulation-based CPR training course within the past 12 months.

Exclusion Criteria:

* Presence of cardiovascular, respiratory, musculoskeletal, or other health conditions that limit the ability to participate in hands-on CPR training.
* Currently experiencing an injury or acute pain that affects the ability to perform chest compressions or other CPR techniques.
* Refusal or withdrawal of consent to participate in the study at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
CPR Skills Performance Score | Baseline (T1), Immediate Post-test (T2), 3-month Follow-up (T3)
  Skills evaluated with a 14-item standardized checklist adapted from American Heart Association guidelines. Includes responsiveness check, EMS activation, breathing assessment, correct hand placement, compression quality, rescue breaths, AED use, and scene safety. Scored 0-14; categorized as poor, needs improvement, competent, or excellent.

SECONDARY OUTCOMES:
CPR Knowledge Score | Baseline (T1), Immediate Post-test (T2), 3-month Follow-up (T3)
  Knowledge assessed using a validated multiple-choice questionnaire adapted from Gao et al. (2024), covering CPR hand position, compression rate, compression-to-ventilation ratio, and cardiac arrest recognition. Items rated on a 5-point Likert scale ("very unclear" to "very clear"); higher scores indicate better knowledge.
Attitude Toward CPR | Baseline (T1), Immediate Post-test (T2), 3-month Follow-up (T3)
  Attitudes measured using an 11-item Likert scale ("strongly disagree" to "strongly agree") assessing beliefs about CPR training value, moral responsibility, and support for public CPR education. Higher scores reflect more positive attitudes.
Self-Efficacy in Performing CPR | Baseline (T1), Immediate Post-test (T2), 3-month Follow-up (T3)
  Self-efficacy measured via a 4-item scale rating confidence in performing chest compressions, rescue breaths, AED use, and scene assessment on a 5-point scale ("not confident at all" to "extremely confident"). Higher scores indicate greater self-efficacy.

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  De-identified individual participant data (IPD) underlying the results reported in this study will be made available to qualified researchers upon reasonable request. The shared dataset will include information on demographic characteristics, primary and secondary outcome measures, and relevant protocol details, excluding any direct identifiers to protect participant confidentiality.
  Time Frame:
  Data will be available beginning 6 months after publication of the primary results and will remain accessible for 5 years thereafter.
  Access Criteria:
  Researchers must submit a methodologically sound proposal, including objectives, study design, and data analysis plan. Requests should be sent to liem.le@eiu.eud.vn. Access will be granted upon review and approval by the principal investigator and the Eastern International University Ethics Committee. Data will be shared via a secure, password-protected repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available starting 6 months after publication of primary results, for up to 5 years.
Access Criteria: Requests must include a methodologically sound proposal and will be reviewed by the principal investigator and the Eastern International University Ethics Committee. Data will be provided via a secure, password-protected repository.